CLINICAL TRIAL: NCT01165229
Title: Efficacy, Safety and Immunogenicity Study of GSK Biologicals' Herpes Zoster Vaccine GSK1437173A in Adults Aged 70 Years or Older
Brief Title: Study to Evaluate Efficacy, Safety and Immunogenicity of GlaxoSmithKline (GSK) Biologicals' Herpes Zoster (HZ) Vaccine GSK1437173A in Adults Aged 70 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 113077; 2009-015791-94 (EudraCT Number)
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Herpes Zoster; Herpes Zoster Vaccine
Keywords: Immunogenicity; Subjects 70 years and older; Efficacy; Herpes Zoster; Safety; Adults; Vaccine
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Zoster vaccine group (Experimental): Subjects will receive Herpes Zoster Vaccine GSK1437173A according to a 0, 2-month schedule
  Interventions: Biological: Herpes Zoster Vaccine GSK1437173A
- Placebo group (Placebo Comparator): Subjects will receive NaCl solution placebo according to a 0, 2-month schedule
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Herpes Zoster Vaccine GSK1437173A — Intramuscular injection
  Arms: Zoster vaccine group
Biological: Placebo — Intramuscular injection.
  Arms: Placebo group

SUMMARY:
The purpose of this observer-blind study is to evaluate the efficacy, safety and immunogenicity of GSK Biologicals' candidate Herpes Zoster (HZ) vaccine in adults aged ≥ 70 years.

Two studies (Zoster-006 [NCT01165177] and Zoster-022 [NCT01165229]) will be conducted concurrently to evaluate efficacy of GSK1437173A vaccine. A pooled analysis of data from both studies combined will be conducted contingent on each study achieving its objectives. This protocol posting also deals with the outcome measures related to the pooled analysis.

DETAILED DESCRIPTION:
This protocol summary has been updated following Protocol Amendment 4 changes to study objectives and endpoints. Pooled analyses of ZOSTER-006 (NCT01165177) and ZOSTER-022 (NCT01165229) will only be conducted if the primary objective herpes zoster vaccine efficacy (HZ VE) is demonstrated in both ZOSTER-006 (NCT01165177) and ZOSTER-022 (NCT01165229) separately.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* A male or female aged 70 years or older at the time of the first vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy History of HZ.
* Previous vaccination against varicella or HZ.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine. Additionally, consider allergic reactions to other material or equipment related to study participation.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study.
* Receipt of immunoglobulins and/or any blood products within the 90 days preceding the first dose of study vaccine or planned administration during the study period.
* Administration or planned administration of any other immunizations within 30 days before the first or second study vaccination or scheduled within 30 days after study vaccination. However, licensed non-replicating vaccines may be administered up to 8 days prior to each dose and/or at least 14 days after any dose of study vaccine.
* Any other condition that, in the opinion of the investigator, might interfere with the evaluations required by the study.
* Acute disease and/or fever at the time of enrolment.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14819 (Actual)
Dates: Start 2010-08-02 (Actual); Primary Completion 2015-07-24 (Actual); Study Completion 2015-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (184):
- United States (39):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Wadsworth, Ohio
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Pleasant Hills, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Arlington, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Winchester, Virginia
  - GSK Investigational Site, Renton, Washington
- Australia (9):
  - GSK Investigational Site, Glebe, New South Wales
  - GSK Investigational Site, Maroubra, New South Wales
  - GSK Investigational Site, Umina, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Wollongong, New South Wales
  - GSK Investigational Site, Caboolture, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Ivanhoe, Victoria
- Brazil (5):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Curitiba/Paraná, Paraná
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Curitiba/PR
  - GSK Investigational Site, São Paulo
- Canada (13):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Woodstock, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, České Budějovice
  - GSK Investigational Site, Hradec Králové
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (9):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- France (13):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Château-Gontier
  - GSK Investigational Site, Cherbourg
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Laval
  - GSK Investigational Site, Montrevault
  - GSK Investigational Site, Muret
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Rosiers-d'Égletons
  - GSK Investigational Site, Saint Cyr Sur Loir
  - GSK Investigational Site, Segré
  - GSK Investigational Site, Soulaines-sur-Aubance
  - GSK Investigational Site, Tours
- Germany (31):
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Güglingen, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Wangen, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Dachau, Bavaria
  - GSK Investigational Site, Künzing, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Rednitzhembach, Bavaria
  - GSK Investigational Site, Wallerfing, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Flörsheim, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Duelmen, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freiberg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Pirna, Saxony
  - GSK Investigational Site, Köthen, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Hong Kong (2):
  - GSK Investigational Site, Kwun Tong
  - GSK Investigational Site, Shatin
- Italy (10):
  - GSK Investigational Site, Chieti, Abruzzo
  - GSK Investigational Site, Pescara, Abruzzo
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Monza, Lombardy
  - GSK Investigational Site, Cuneo, Piedmont
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Ragusa (RG), Sicily
- Japan (4):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Tokyo
- Mexico (4):
  - GSK Investigational Site, Zapopan, Jalisco, Jalisco
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, Durango
  - GSK Investigational Site, Monterrey
- South Korea (6):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Kangnam-gu, Seoul
  - GSK Investigational Site, Kangwon-do
  - GSK Investigational Site, Seoul
- Spain (10):
  - GSK Investigational Site, Alcover( Tarragona)
  - GSK Investigational Site, Balenyà (Barcelona)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Centelles
  - GSK Investigational Site, La Roca Del Valles (Barcelona)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda
  - GSK Investigational Site, Peralada( Girona)
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vic/ Barcelona
- Sweden (12):
  - GSK Investigational Site, Borås
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Jönköping
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Skövde
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
  - GSK Investigational Site, Vällingby
- Taiwan (3):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- United Kingdom (9):
  - GSK Investigational Site, Buckshaw Village, Chorley, Lancashire
  - GSK Investigational Site, Atherstone, Warwickshire
  - GSK Investigational Site, Bradford-on-Avon, Wiltshire
  - GSK Investigational Site, Bangor
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Broughshane
  - GSK Investigational Site, Ledbury
  - GSK Investigational Site, Newtonabbey
  - GSK Investigational Site, Waterloo, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Background] Cunningham AL, Lal H, Kovac M, Chlibek R, Hwang SJ, Diez-Domingo J, Godeaux O, Levin MJ, McElhaney JE, Puig-Barbera J, Vanden Abeele C, Vesikari T, Watanabe D, Zahaf T, Ahonen A, Athan E, Barba-Gomez JF, Campora L, de Looze F, Downey HJ, Ghesquiere W, Gorfinkel I, Korhonen T, Leung E, McNeil SA, Oostvogels L, Rombo L, Smetana J, Weckx L, Yeo W, Heineman TC; ZOE-70 Study Group. Efficacy of the Herpes Zoster Subunit Vaccine in Adults 70 Years of Age or Older. N Engl J Med. 2016 Sep 15;375(11):1019-32. doi: 10.1056/NEJMoa1603800. PMID 27626517
- [Background] Cunningham AL, Heineman TC, Lal H, Godeaux O, Chlibek R, Hwang SJ, McElhaney JE, Vesikari T, Andrews C, Choi WS, Esen M, Ikematsu H, Choma MK, Pauksens K, Ravault S, Salaun B, Schwarz TF, Smetana J, Abeele CV, Van den Steen P, Vastiau I, Weckx LY, Levin MJ; ZOE-50/70 Study Group. Immune Responses to a Recombinant Glycoprotein E Herpes Zoster Vaccine in Adults Aged 50 Years or Older. J Infect Dis. 2018 May 5;217(11):1750-1760. doi: 10.1093/infdis/jiy095. PMID 29529222
- [Background] Ikematsu H et al. (2018) Efficacy, safety and immunogenicity of new adjuvanted herpes zoster subunit vaccine for Japanese over 50 years old and over 70 years old. Kansenshogaku Zasshi. 92(2):103-114.
- [Background] Kovac M, Lal H, Cunningham AL, Levin MJ, Johnson RW, Campora L, Volpi A, Heineman TC; ZOE-50/70 Study Group. Complications of herpes zoster in immunocompetent older adults: Incidence in vaccine and placebo groups in two large phase 3 trials. Vaccine. 2018 Mar 14;36(12):1537-1541. doi: 10.1016/j.vaccine.2018.02.029. Epub 2018 Feb 17. PMID 29463421
- [Derived] Matthews S, Curran D, Sabater Cabrera E, Boutry C, Lecrenier N, Cunningham AL, Schmader K. An Analysis of How Herpes Zoster Pain Affects Health-related Quality of Life of Placebo Patients From 3 Randomized Phase III Studies. Clin J Pain. 2023 Aug 1;39(8):386-393. doi: 10.1097/AJP.0000000000001129. PMID 37166199
- [Derived] Kim JH, Johnson R, Kovac M, Cunningham AL, Amakrane M, Sullivan KM, Dagnew AF, Curran D, Schuind A. Adjuvanted recombinant zoster vaccine decreases herpes zoster-associated pain and the use of pain medication across 3 randomized, placebo-controlled trials. Pain. 2023 Apr 1;164(4):741-748. doi: 10.1097/j.pain.0000000000002760. Epub 2022 Aug 19. PMID 36066965
- [Derived] Kim JH, Diaz-Decaro J, Jiang N, Hwang SJ, Choo EJ, Co M, Hastie A, Hui DSC, Irimajiri J, Lee J, Leung EM, Tang H, Tsuru T, Watson P, Wu Z, Yu CJ, Yuan Y, Zahaf T, Cunningham AL, Schuind A. The adjuvanted recombinant zoster vaccine is efficacious and safe in Asian adults >/= 50 years of age: a sub-cohort analysis of the ZOE-50 and ZOE-70 randomized trials. Hum Vaccin Immunother. 2021 Jul 3;17(7):2050-2057. doi: 10.1080/21645515.2020.1859321. Epub 2021 Feb 19. PMID 33606577
- [Derived] Dagnew AF, Rausch D, Herve C, Zahaf T, Levin MJ, Schuind A; ZOE-50/70 study group. Efficacy and serious adverse events profile of the adjuvanted recombinant zoster vaccine in adults with pre-existing potential immune-mediated diseases: a pooled post hoc analysis on two parallel randomized trials. Rheumatology (Oxford). 2021 Mar 2;60(3):1226-1233. doi: 10.1093/rheumatology/keaa424. PMID 32910152
- [Derived] Colindres R, Wascotte V, Brecx A, Clarke C, Herve C, Kim JH, Levin MJ, Oostvogels L, Zahaf T, Schuind A, Cunningham AL. Post hoc analysis of reactogenicity trends between dose 1 and dose 2 of the adjuvanted recombinant zoster vaccine in two parallel randomized trials. Hum Vaccin Immunother. 2020 Nov 1;16(11):2628-2633. doi: 10.1080/21645515.2020.1741312. Epub 2020 Apr 29. PMID 32347767
- [Derived] Willer DO, Oostvogels L, Cunningham AL, Gervais P, Gorfinkel I, Hyung Kim J, Talarico C, Wascotte V, Zahaf T, Colindres R, Schuind A; ZOE 50/70 study groups. Efficacy of the adjuvanted recombinant zoster vaccine (RZV) by sex, geographic region, and geographic ancestry/ethnicity: A post-hoc analysis of the ZOE-50 and ZOE-70 randomized trials. Vaccine. 2019 Oct 8;37(43):6262-6267. doi: 10.1016/j.vaccine.2019.09.028. Epub 2019 Sep 16. PMID 31537443
- [Derived] Lopez-Fauqued M, Campora L, Delannois F, El Idrissi M, Oostvogels L, De Looze FJ, Diez-Domingo J, Heineman TC, Lal H, McElhaney JE, McNeil SA, Yeo W, Tavares-Da-Silva F; ZOE-50/70 Study Group. Safety profile of the adjuvanted recombinant zoster vaccine: Pooled analysis of two large randomised phase 3 trials. Vaccine. 2019 Apr 24;37(18):2482-2493. doi: 10.1016/j.vaccine.2019.03.043. Epub 2019 Mar 29. PMID 30935742
- [Derived] Curran D, Oostvogels L, Heineman T, Matthews S, McElhaney J, McNeil S, Diez-Domingo J, Lal H, Andrews C, Athan E, Berglund J, Campora L, de Looze F, Korhonen T, Leung E, Levin M, Volpi A, Johnson RW; ZOE-50/70 Study Group. Quality of Life Impact of an Adjuvanted Recombinant Zoster Vaccine in Adults Aged 50 Years and Older. J Gerontol A Biol Sci Med Sci. 2019 Jul 12;74(8):1231-1238. doi: 10.1093/gerona/gly150. PMID 29955836
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 13900 subjects from the total enrolled number were vaccinated and included in the Total Vaccinated Cohort. In the placebo group,1 subject had an unknown withdrawal status before the study site closure. This was not identified during database freeze, leading to 1190 subjects in place of 1189 that actually completed the placebo group
Groups:
- Zoster-022 GSK1437173A Group: Subjects receiving herpes zoster subunit vaccine (gE/AS01B vaccine) according to a 0, 2-month schedule.
- Zoster-022 Placebo Group: Subjects receiving saline solution (NaCl solution) as control according to a 0, 2-month schedule.
Period: Overall Study
Arm/Group | Zoster-022 GSK1437173A Group | Zoster-022 Placebo Group
Started | 6950 | 6950
Completed | 5770 | 5760
Not Completed | 1180 | 1190
Not completed — Serious Adverse Event | 456 | 487
Not completed — Non-Serious Adverse Event | 47 | 15
Not completed — Protocol Violation | 6 | 8
Not completed — Withdrawal by Subject | 387 | 396
Not completed — Migrated/moved from study area | 51 | 46
Not completed — Lost to Follow-up | 123 | 133
Not completed — Suspected HZ Episode | 2 | 2
Not completed — No reason from the subject | 108 | 102
Not completed — Unknown completion status | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoster-022 GSK1437173A Group | Zoster-022 Placebo Group | Total
Number analyzed (Participants) | 6950 | 6950 | 13900
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.6 (4.7) | 75.6 (4.7) | 75.6 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3789 | 3836 | 7625
  Male | 3161 | 3114 | 6275
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African Heritage / African American | 79 | 67 | 146
  Geographic ancestry: American Indian or Alaskan Native | 1 | 8 | 9
  Geographic ancestry: Asian - Central/South Asian Heritage | 3 | 6 | 9
  Geographic ancestry: Asian - East Asian Heritage | 907 | 908 | 1815
  Geographic ancestry: Asian - Japanese Heritage | 298 | 300 | 598
  Geographic ancestry: Asian - South East Asian Heritage | 8 | 4 | 12
  Geographic ancestry: Native Hawaiian or Other Pacific Islander | 3 | 3 | 6
  Geographic ancestry: White - Arabic / North African Heritage | 40 | 47 | 87
  Geographic ancestry: White - Caucasian / European Heritage | 5307 | 5301 | 10608
  Geographic ancestry: Other | 304 | 306 | 610

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Episodes of Herpes Zoster (HZ)
Description: Confirmed HZ cases during the study in the modified total vaccinated cohort (mTVc).
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: The analysis was based on the modified total vaccinated cohort, which included subjects from the total vaccinated cohort, except those who were not administered with the second vaccination or who developed a confirmed case of Herpes Zoster prior to 1 month after the second vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Zoster-022 GSK1437173A 70-79YOA Group: Subjects between 70 and 79 years of age (YOA), receiving herpes zoster subunit vaccine (gE/AS01B vaccine) according to a 0, 2-month schedule.
- Zoster-022 GSK1437173A >=80YOA Group: Subjects above 80 years of age (YOA), receiving herpes zoster subunit vaccine (gE/AS01B vaccine) according to a 0, 2-month schedule.
- Zoster-022 GSK1437173A >=70YOA Group: Subjects above 70 years of age (YOA), receiving herpes zoster subunit vaccine (gE/AS01B vaccine) according to a 0, 2-month schedule.
- Zoster-022 Placebo 70-79YOA Group: Subjects between 70 and 79 years of age (YOA), receiving saline solution (NaCl solution) as control according to a 0, 2-month schedule.
- Zoster-022 Placebo >=80YOA Group: Subjects above 80 years of age (YOA), receiving saline solution (NaCl solution) as control according to a 0, 2-month schedule.
- Zoster-022 Placebo >=70YOA Group: Subjects above 70 years of age (YOA), receiving saline solution (NaCl solution) as control according to a 0, 2-month schedule.
Arm/Group | Zoster-022 GSK1437173A 70-79YOA Group | Zoster-022 GSK1437173A >=80YOA Group | Zoster-022 GSK1437173A >=70YOA Group | Zoster-022 Placebo 70-79YOA Group | Zoster-022 Placebo >=80YOA Group | Zoster-022 Placebo >=70YOA Group
Number analyzed (Participants) | 5114 | 1427 | 6541 | 5189 | 1433 | 6622
Participants | 17 | 6 | 23 | 169 | 54 | 223
Statistical Analysis 1: Comparison: Zoster-022 GSK1437173A 70-79YOA Group vs Zoster-022 Placebo 70-79YOA Group; Comparison of vaccine efficacy in prevention of Herpes Zoster (HZ) disease between Zoster-022 GSK1437173A 70-79 YOA group and Zoster-022 Placebo 70-79 YOA group; Test type: Other — The efficacy of Herpes Zoster subunit (HZ/su) vaccine against herpes zoster disease was demonstrated if the lower limit (LL) of the two-sided 95% Confidence Interval (CI) of VE was above 10%; p < 0.0001, Poisson exact test; Vaccine efficacy = 90.02, 95% CI 2-sided [83.54 to 94.32]
Statistical Analysis 2: Comparison: Zoster-022 GSK1437173A >=80YOA Group vs Zoster-022 Placebo >=80YOA Group; Comparison of vaccine efficacy in prevention of Herpes Zoster (HZ) disease between Zoster-022 GSK1437173A >=80YOA Group and Zoster-022 Placebo Zoster-022 Placebo >=80YOA Group; Test type: Other — The efficacy of HZ/su vaccine against herpes zoster disease was demonstrated if the lower limit of the of the 2-sided 95% CI of VE was above 10%; p < 0.0001, Poisson exact method; Vaccine efficacy = 89.08, 95% CI 2-sided [74.65 to 96.16]
Statistical Analysis 3: Comparison: Zoster-022 GSK1437173A >=70YOA Group vs Zoster-022 Placebo >=70YOA Group; Comparison of vaccine efficacy in prevention of Herpes Zoster (HZ) disease between Zoster-022 GSK1437173A >=70YOA Group and Zoster-022 Placebo >=70YOA Group; Test type: Other — [test comment as in outcome 1, analysis 2]; p < 0.0001, Poisson exact test; Vaccine efficacy = 89.79, 95% CI 2-sided [84.29 to 93.66]

2. Primary Outcome: Outcome Measure for the Pooled Analysis of Combined Data From Studies ZOSTER-006 (NCT01165177) and ZOSTER-022 (NCT01165229): Number of Subjects With Post-herpetic Neuralgia (PHN)
Description: Incidence of PHN calculated using the mTVc during the entire study period in subjects ≥ 70 years of age (YOA).
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Zoster-022/006 Pooled GSK1437173A 70-79YOA Group: Subjects between 70 and 79 years of age (YOA), receiving herpes zoster subunit vaccine (gE/AS01B vaccine) according to a 0, 2-month schedule.
- Zoster-022/006 Pooled GSK1437173A >=80YOA Group: Subjects above 80 years of age (YOA), receiving herpes zoster subunit vaccine (gE/AS01B vaccine) according to a 0, 2-month schedule.
- Zoster-022/006 Pooled GSK1437173A >=70YOA Group: Subjects above 70 years of age (YOA), receiving herpes zoster subunit vaccine (gE/AS01B vaccine) according to a 0, 2-month schedule.
- Zoster-022/006 Pooled Placebo 70-79YOA Group: Subjects between 70 and 79 years of age (YOA), receiving saline solution (NaCl solution) as control according to a 0, 2-month schedule.
- Zoster-022/006 Pooled Placebo >=80YOA Group: Subjects above 80 years of age (YOA), receiving saline solution (NaCl solution) as control according to a 0, 2-month schedule.
- Zoster-022/006 Pooled Placebo >=70YOA Group: Subjects above 70 years of age (YOA), receiving saline solution (NaCl solution) as control according to a 0, 2-month schedule.
Arm/Group | Zoster-022/006 Pooled GSK1437173A 70-79YOA Group | Zoster-022/006 Pooled GSK1437173A >=80YOA Group | Zoster-022/006 Pooled GSK1437173A >=70YOA Group | Zoster-022/006 Pooled Placebo 70-79YOA Group | Zoster-022/006 Pooled Placebo >=80YOA Group | Zoster-022/006 Pooled Placebo >=70YOA Group
Number analyzed (Participants) | 6468 | 1782 | 8250 | 6554 | 1792 | 8346
Participants | 2 | 2 | 4 | 29 | 7 | 36
Statistical Analysis 1: Comparison: Zoster-022/006 Pooled GSK1437173A 70-79YOA Group vs Zoster-022/006 Pooled Placebo 70-79YOA Group; Comparison of vaccine efficacy in prevention of Post-Herpetic Neuralgia (PHN) between Zoster-022/006 Pooled GSK1437173A 70-79YOA Group and Zoster-022/006 Pooled Placebo 70-79YOA Group; Test type: Other — The efficacy of HZ/su vaccine against PHN was demonstrated if the lower limit of the of the 2-sided 95% CI of VE was above 0%; p < 0.0001, Poisson exact test; Vaccine efficacy = 93.04, 95% CI 2-sided [72.47 to 99.19]
Statistical Analysis 2: Comparison: Zoster-022/006 Pooled GSK1437173A >=80YOA Group vs Zoster-022/006 Pooled Placebo >=80YOA Group; Comparison of vaccine efficacy in prevention of PHN between Zoster-022/006 Pooled GSK1437173A >=80YOA Group and Zoster-022/006 Pooled Placebo >=80YOA Group; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.1844, Poisson exact test; Vaccine efficacy = 71.16, 95% CI 2-sided [-51.51 to 97.08]
Statistical Analysis 3: Comparison: Zoster-022/006 Pooled GSK1437173A >=70YOA Group vs Zoster-022/006 Pooled Placebo >=70YOA Group; Comparison of vaccine efficacy in prevention of PHN between Zoster-022/006 Pooled GSK1437173A >=70YOA Group and Zoster-022/006 Pooled Placebo >=70YOA Group; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, Poisson exact test; Vaccine efficacy = 88.78, 95% CI 2-sided [68.70 to 97.10]

3. Primary Outcome: Outcome Measure for the Pooled Analysis of Combined Data From Studies Zoster-006 (NCT01165177) and Zoster-022 (NCT01165229): Number of Subjects With Confirmed HZ
Description: Occurrence of confirmed HZ during the entire study period in subjects ≥ 70 YOA.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022/006 Pooled GSK1437173A 70-79YOA Group | Zoster-022/006 Pooled GSK1437173A >=80YOA Group | Zoster-022/006 Pooled GSK1437173A >=70YOA Group | Zoster-022/006 Pooled Placebo 70-79YOA Group | Zoster-022/006 Pooled Placebo >=80YOA Group | Zoster-022/006 Pooled Placebo >=70YOA Group
Number analyzed (Participants) | 6468 | 1782 | 8250 | 6554 | 1792 | 8346
Participants | 19 | 6 | 25 | 216 | 68 | 284
Statistical Analysis 1: Comparison: Zoster-022/006 Pooled GSK1437173A 70-79YOA Group vs Zoster-022/006 Pooled Placebo 70-79YOA Group; Comparison of vaccine efficacy in prevention of herpes zoster disease between Zoster-022/006 Pooled GSK1437173A 70-79YOA Group and Zoster-022/006 Pooled Placebo 70-79YOA Group; Test type: Other — [test comment as in outcome 1, analysis 2]; p < 0.0001, Poisson exact test; Vaccine efficacy = 91.27, 95% CI 2-sided [86.04 to 94.85]
Statistical Analysis 2: Comparison: Zoster-022/006 Pooled GSK1437173A >=80YOA Group vs Zoster-022/006 Pooled Placebo >=80YOA Group; Comparison of vaccine efficacy in prevention of herpes zoster disease between Zoster-022/006 Pooled GSK1437173A >=80YOA Group and Zoster-022/006 Pooled Placebo >=80YOA Group; Test type: Other — [test comment as in outcome 1, analysis 2]; p < 0.0001, Poisson exact test; Vaccine efficacy = 91.37, 95% CI 2-sided [80.22 to 96.94]
Statistical Analysis 3: Comparison: Zoster-022/006 Pooled GSK1437173A >=70YOA Group vs Zoster-022/006 Pooled Placebo >=70YOA Group; Comparison of vaccine efficacy in prevention of herpes zoster disease between Zoster-022/006 pooled GSK1437173A >=70 YOA Group and Zoster-022/006 Pooled Placebo >=70YOA Group; Test type: Other — [test comment as in outcome 1, analysis 2]; p < 0.0001, Poisson exact test; Vaccine efficacy = 91.30, 95% CI 2-sided [86.88 to 94.46]

4. Secondary Outcome: Number of Subjects With Post-herpetic Neuralgia (PHN)
Description: PHN cases in the mTVc.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022 GSK1437173A 70-79YOA Group | Zoster-022 GSK1437173A >=80YOA Group | Zoster-022 GSK1437173A >=70YOA Group | Zoster-022 Placebo 70-79YOA Group | Zoster-022 Placebo >=80YOA Group | Zoster-022 Placebo >=70YOA Group
Number analyzed (Participants) | 5114 | 1427 | 6541 | 5189 | 1433 | 6622
Participants | 2 | 2 | 4 | 22 | 6 | 28
Statistical Analysis 1: Comparison: Zoster-022 GSK1437173A 70-79YOA Group vs Zoster-022 Placebo 70-79YOA Group; Comparison of of Vaccine Efficacy (VE) in prevention of PHN between Zoster-022 GSK1437173A 70-79YOA Group and Zoster-022 placebo 70-79YOA Group; Test type: Other — The efficacy of HZ/su vaccine against PHN was demonstrated if the LL of the two-sided 95% CI of VE was above 0%; p < 0.0001, Poisson exact test; Vaccine efficacy = 90.80, 95% CI 2-sided [62.57 to 98.95]
Statistical Analysis 2: Comparison: Zoster-022 GSK1437173A >=80YOA Group vs Zoster-022 Placebo >=80YOA Group; Comparison of vaccine efficacy in prevention of PHN between Zoster-022 GSK1437173A >=80YOA Group and Zoster-022 Placebo >=80YOA Group; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.3072, Poisson exact test; Vaccine efficacy = 65.76, 95% CI 2-sided [-91.58 to 96.62]
Statistical Analysis 3: Comparison: Zoster-022 GSK1437173A >=70YOA Group vs Zoster-022 Placebo >=70YOA Group; Comparison of vaccine efficacy in prevention of PHN between Zoster-022 GSK1437173A >=70YOA Group and Zoster-022 Placebo >=70YOA Group; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, Poisson exact test; Vaccine efficacy = 85.49, 95% CI 2-sided [58.52 to 96.30]

5. Secondary Outcome: Number of Days With Severe 'Worst' HZ-associated Pain
Description: Duration of severe 'worst' HZ-associated pain following the onset of a confirmed HZ rash over the entire pain reporting period as measured by the Zoster Brief Pain Inventory (ZBPI) in subjects with confirmed HZ.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Zoster-022 GSK1437173A 70-79YOA Group | Zoster-022 GSK1437173A >=80YOA Group | Zoster-022 GSK1437173A >=70YOA Group | Zoster-022 Placebo 70-79YOA Group | Zoster-022 Placebo >=80YOA Group | Zoster-022 Placebo >=70YOA Group
Number analyzed (Participants) | 15 | 3 | 18 | 150 | 48 | 198
Days | 21.8 (31.41) | 98.7 (57.73) | 34.6 (45.54) | 47.9 (100.08) | 50.4 (106.51) | 48.5 (101.40)
Statistical Analysis 1: Comparison: Zoster-022 GSK1437173A 70-79YOA Group vs Zoster-022 Placebo 70-79YOA Group; Comparison of VE in reduction of duration of severe worst HZ associated pain between Zoster-022 GSK1437173A 70-79YOA Group and Zoster-022 Placebo 70-79YOA Group; Test type: Other — The efficacy of HZ/su vaccine against duration of severe worst HZ associated pain was demonstrated if the LL of the two-sided 95% CI of VE derived from the Hazard ratio was above 0%; p = 0.3749, Poisson exact test; Vaccine efficacy = 21.70, 95% CI 2-sided [-34.40 to 54.39]
Statistical Analysis 2: Comparison: Zoster-022 GSK1437173A >=80YOA Group vs Zoster-022 Placebo >=80YOA Group; Comparison of VE in reduction of duration of severe worst HZ associated pain between Zoster-022 GSK1437173A >=80YOA Group and Zoster-022 Placebo>=80YOA Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.2466, Poisson exact test; Vaccine efficacy = 51.76, 95% CI 2-sided [-65.55 to 85.95]
Statistical Analysis 3: Comparison: Zoster-022 GSK1437173A >=70YOA Group vs Zoster-022 Placebo >=70YOA Group; Comparison of VE in reduction of duration of severe worst HZ associated pain between Zoster-022 GSK1437173A >=70YOA Group and Zoster-022 Placebo>=70YOA Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.1877, Poisson exact test; Vaccine efficacy = 28.40, 95% CI 2-sided [-17.69 to 56.44]

6. Secondary Outcome: Number of Subjects With Confirmed HZ Episode Related Mortality and Hospitalizations
Description: The number of subjects with confirmed HZ related mortality and hospitalizations were tabulated.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022 GSK1437173A 70-79YOA Group | Zoster-022 GSK1437173A >=80YOA Group | Zoster-022 GSK1437173A >=70YOA Group | Zoster-022 Placebo 70-79YOA Group | Zoster-022 Placebo >=80YOA Group | Zoster-022 Placebo >=70YOA Group
Number analyzed (Participants) | 5114 | 1427 | 6541 | 5189 | 1433 | 6622
Participants
  Mortality | 0 | 0 | 0 | 0 | 0 | 0
  Hospitalization | 0 | 0 | 0 | 3 | 2 | 5
  Mortality or hospitalization | 0 | 0 | 0 | 3 | 2 | 5

7. Secondary Outcome: Number of Subjects With Overall Mortality and HZ-related Mortality
Description: The number of subjects with overall mortality and HZ related mortality were tabulated. Evaluation of VE in the reduction of overall and HZ related mortality as per study objective was not performed due to low number of events reported.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022 GSK1437173A 70-79YOA Group | Zoster-022 GSK1437173A >=80YOA Group | Zoster-022 GSK1437173A >=70YOA Group | Zoster-022 Placebo 70-79YOA Group | Zoster-022 Placebo >=80YOA Group | Zoster-022 Placebo >=70YOA Group
Number analyzed (Participants) | 5114 | 1427 | 6541 | 5189 | 1433 | 6622
Participants | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Subjects With Confirmed HZ Episode Related Hospitalizations
Description: Incidence of overall and HZ-related hospitalizations during the study.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022 GSK1437173A 70-79YOA Group | Zoster-022 GSK1437173A >=80YOA Group | Zoster-022 GSK1437173A >=70YOA Group | Zoster-022 Placebo 70-79YOA Group | Zoster-022 Placebo >=80YOA Group | Zoster-022 Placebo >=70YOA Group
Number analyzed (Participants) | 5114 | 1427 | 6541 | 5189 | 1433 | 6622
Participants | 0 | 0 | 0 | 3 | 2 | 5
Statistical Analysis 1: Comparison: Zoster-022 GSK1437173A 70-79YOA Group vs Zoster-022 Placebo 70-79YOA Group; Comparison of VE in reduction of overall and HZ related hospitalizations between Zoster-022 GSK1437173A 70-79YOA Group and Zoster-022 Placebo 70-79YOA Group; Test type: Other — Efficacy of the HZ/su vaccine against overall and HZ related hospitalizations was demonstrated if the LL of the two-sided 95% CI of VE was above 0%; p = 0.2533, Poisson exact test; Vaccine efficacy = 100.00, 95% CI 2-sided [-144.13 to 100.00]
Statistical Analysis 2: Comparison: Zoster-022 GSK1437173A >=80YOA Group vs Zoster-022 Placebo >=80YOA Group; Comparison of VE in reduction of overall and HZ related hospitalizations between Zoster-022 GSK1437173A >=80YOA Group and Zoster-022 Placebo >=80YOA Group; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.5024, Poisson exact test; Vaccine efficacy = 100.00, 95% CI 2-sided [-435.14 to 100.00]
Statistical Analysis 3: Comparison: Zoster-022 GSK1437173A >=70YOA Group vs Zoster-022 Placebo >=70YOA Group; Comparison of VE in reduction of overall and HZ related hospitalizations between Zoster-022 GSK1437173A >=70YOA Group and Zoster-022 Placebo >=70YOA Group; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.0636, Poisson exact test; Vaccine efficacy = 100.00, 95% CI 2-sided [-9.92 to 100.00]

9. Secondary Outcome: Number of Subjects With HZ Related Complications
Description: Incidence of HZ complications during the study in subjects with confirmed HZ.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022 GSK1437173A 70-79YOA Group | Zoster-022 GSK1437173A >=80YOA Group | Zoster-022 GSK1437173A >=70YOA Group | Zoster-022 Placebo 70-79YOA Group | Zoster-022 Placebo >=80YOA Group | Zoster-022 Placebo >=70YOA Group
Number analyzed (Participants) | 17 | 6 | 23 | 169 | 54 | 223
Participants
  At least one complication | 1 | 0 | 1 | 6 | 4 | 10
  HZ vasculitis | 0 | 0 | 0 | 0 | 0 | 0
  Disseminated Disease | 0 | 0 | 0 | 0 | 2 | 2
  Ophthalmic Disease | 1 | 0 | 1 | 4 | 2 | 6
  Neurologic Disease | 0 | 0 | 0 | 3 | 0 | 3
  Visceral Disease | 0 | 0 | 0 | 0 | 0 | 0
  Stroke | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Zoster-022 GSK1437173A 70-79YOA Group vs Zoster-022 Placebo 70-79YOA Group; Comparison of VE in reduction of HZ related complications between Zoster-022 GSK1437173A 70-79YOA Group and Zoster-022 Placebo 70-79YOA Group; Test type: Other — Efficacy of the HZ/su vaccine against HZ related complications was demonstrated if the LL of the VE was above 0%; p = 0.4947, Poisson exact test; Vaccine efficacy = -65.69, 95% CI 2-sided [-827.06 to 73.62]
Statistical Analysis 2: Comparison: Zoster-022 GSK1437173A >=80YOA Group vs Zoster-022 Placebo >=80YOA Group; Comparison of VE in reduction of HZ related complications between Zoster-022 GSK1437173A >=80YOA Group and Zoster-022 Placebo >=80YOA Group; Test type: Other — Efficacy of the HZ/su vaccine against HZ related complications was demonstrated if the LL of the VE was above 0%; p = 1.0000, Poisson exact test; Vaccine efficacy = 100.00, 95% CI 2-sided [-558.05 to 100.00]
Statistical Analysis 3: Comparison: Zoster-022 GSK1437173A >=70YOA Group vs Zoster-022 Placebo >=70YOA Group; Comparison of VE in reduction of HZ related complications between Zoster-022 GSK1437173A >=70YOA Group and Zoster-022 Placebo >=70YOA Group; Test type: Other — Efficacy of the HZ/su vaccine against HZ related complications was demonstrated if the LL of the VE was above 0%; p = 1.0000, Poisson exact test; Vaccine efficacy = 0.97, 95% CI 2-sided [-433.32 to 83.16]

10. Secondary Outcome: Number of Subjects Receiving Pain Medication Associated With HZ
Description: Incidence of use of pain medications throughout the study
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022 GSK1437173A 70-79YOA Group | Zoster-022 GSK1437173A >=80YOA Group | Zoster-022 GSK1437173A >=70YOA Group | Zoster-022 Placebo 70-79YOA Group | Zoster-022 Placebo >=80YOA Group | Zoster-022 Placebo >=70YOA Group
Number analyzed (Participants) | 17 | 6 | 23 | 169 | 54 | 223
Participants
  At least 1 pain medication | 7 | 3 | 10 | 123 | 37 | 160
  1 pain medication only | 5 | 0 | 5 | 43 | 17 | 60
  2 pain medications only | 0 | 1 | 1 | 30 | 4 | 34
  3 pain medications or more | 2 | 2 | 4 | 50 | 16 | 66
Statistical Analysis 1: Comparison: Zoster-022 GSK1437173A 70-79YOA Group vs Zoster-022 Placebo 70-79YOA Group; Comparison of VE in reduction in use of pain medication between Zoster-022 GSK1437173A 70-79YOA Group and Zoster-022 Placebo 70-79YOA Group; Test type: Other — Efficacy of the HZ/su vaccine against use of pain medications was demonstrated if the LL of the two-sided 95% CI of VE was above 0%; p = 0.0112, Poisson exact test; Vaccine efficacy = 43.42, 95% CI 2-sided [10.77 to 70.53]
Statistical Analysis 2: Comparison: Zoster-022 GSK1437173A >=80YOA Group vs Zoster-022 Placebo >=80YOA Group; Comparison of VE in reduction in use of pain medication between Zoster-022 GSK1437173A >=80YOA Group and Zoster-022 Placebo >=80YOA Group; Test type: Other — Efficacy of the HZ/su vaccine against use of pain medications was demonstrated if the LL of the two-sided 95% CI of the VE was above 0%; p = 0.3903, Poisson exact test; Vaccine efficacy = 27.03, 95% CI 2-sided [-26.43 to 73.20]
Statistical Analysis 3: Comparison: Zoster-022 GSK1437173A >=70YOA Group vs Zoster-022 Placebo >=70YOA Group; Comparison of VE in reduction in use of pain medication between Zoster-022 GSK1437173A >=70YOA group and Zoster-022 Placebo >=70YOA Group; Test type: Other — [test comment as in outcome 10, analysis 1]; p = 0.0083, Poisson exact test; Vaccine efficacy = 39.60, 95% CI 2-sided [10.79 to 64.75]

11. Secondary Outcome: Number of Days With Pain Medication Associated With HZ
Description: Incidence of reduction of duration of pain medication associated with HZ throughout the study.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Zoster-022 GSK1437173A 70-79YOA Group | Zoster-022 GSK1437173A >=80YOA Group | Zoster-022 GSK1437173A >=70YOA Group | Zoster-022 Placebo 70-79YOA Group | Zoster-022 Placebo >=80YOA Group | Zoster-022 Placebo >=70YOA Group
Number analyzed (Participants) | 7 | 3 | 10 | 123 | 37 | 160
Days | 38.7 (56.44) | 274.7 (337.00) | 109.5 (200.88) | 218.6 (593.80) | 135.0 (207.31) | 199.3 (530.60)
Statistical Analysis 1: Comparison: Zoster-022 GSK1437173A 70-79YOA Group vs Zoster-022 Placebo 70-79YOA Group; Comparison of VE in reduction in duration of pain medication associated with HZ between Zoster-022 GSK1437173A 70-79YOA Group and Zoster-022 Placebo 70-79YOA Group; Test type: Other — Efficacy of the HZ/su vaccine against duration of pain medication associated with HZ was demonstrated if the LL of the two-sided 95% CI of VE derived from the hazard ratio was above 0%; p = 0.0232, Poisson exact test; Vaccine efficacy = 58.94, 95% CI 2-sided [11.45 to 80.96]
Statistical Analysis 2: Comparison: Zoster-022 GSK1437173A >=80YOA Group vs Zoster-022 Placebo >=80YOA Group; Comparison of VE in reduction in duration of pain medication associated with HZ between Zoster-022 GSK1437173A >=80YOA Group and Zoster-022 Placebo >=80YOA Group; Test type: Other — [test comment as in outcome 11, analysis 1]; p = 0.8324, Poisson exact test; Vaccine efficacy = -14.56, 95% CI 2-sided [-303.30 to 67.46]
Statistical Analysis 3: Comparison: Zoster-022 GSK1437173A >=70YOA Group vs Zoster-022 Placebo >=70YOA Group; Comparison of VE in reduction in duration of pain medication associated with HZ between Zoster-022 GSK1437173A >=70YOA Group and Zoster-022 Placebo >=70YOA Group; Test type: Other — [test comment as in outcome 11, analysis 1]; p = 0.0404, Poisson exact test; Vaccine efficacy = 49.25, 95% CI 2-sided [2.92 to 73.47]

12. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Occurrence, intensity of each solicited local symptom within 7 days (Days 0-6) after each vaccination, in subjects included in the 7-day diary card subset; Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = Significant pain at rest that prevented everyday normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: Within the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the total vaccinated cohort - Diary Card, which was a subset of subjects from the total vaccinated cohort, who completed diary cards with any solicited symptoms during the 7 days (Day 0 to Day 6) post vaccination period
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022 GSK1437173A Group | Zoster-022 Placebo Group
Number analyzed (Participants) | 505 | 505
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 502 | 504
  Any Pain, Dose 1 | 297 | 26
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 502 | 504
  Grade 3 Pain, Dose 1 | 12 | 1
  Any Redness, Dose 1: number analyzed (Participants) | 502 | 504
  Any Redness, Dose 1 | 143 | 3
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 502 | 504
  Grade 3 Redness, Dose 1 | 9 | 0
  Any Swelling, Dose 1: number analyzed (Participants) | 502 | 504
  Any Swelling, Dose 1 | 85 | 2
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 502 | 504
  Grade 3 Swelling, Dose 1 | 2 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 492 | 491
  Any Pain, Dose 2 | 282 | 23
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 492 | 491
  Grade 3 Pain, Dose 2 | 12 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 492 | 491
  Any Redness, Dose 2 | 137 | 3
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 492 | 491
  Grade 3 Redness, Dose 2 | 15 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 492 | 491
  Any Swelling, Dose 2 | 68 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 492 | 491
  Grade 3 Swelling, Dose 2 | 7 | 0
  Any Pain, Across Doses | 347 | 43
  Grade 3 Pain, Across Doses | 22 | 1
  Any Redness, Across Doses | 198 | 5
  Grade 3 Redness, Across Doses | 20 | 0
  Any Swelling, Across Doses | 114 | 2
  Grade 3 Swelling, Across Doses | 8 | 0

13. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms (including nausea, vomiting, diarrhea and/or abdominal pain), headache, myalgia, shivering and fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022 GSK1437173A Group | Zoster-022 Placebo Group
Number analyzed (Participants) | 504 | 505
Participants
  Any Fatigue, Dose 1: number analyzed (Participants) | 501 | 503
  Any Fatigue, Dose 1 | 104 | 56
  Grade 3 Fatigue, Dose 1: number analyzed (Participants) | 501 | 503
  Grade 3 Fatigue, Dose 1 | 8 | 4
  Related Fatigue, Dose 1: number analyzed (Participants) | 501 | 503
  Related Fatigue, Dose 1 | 85 | 34
  Any Gastrointestinal, Dose 1: number analyzed (Participants) | 501 | 503
  Any Gastrointestinal, Dose 1 | 25 | 28
  Grade 3 Gastrointestinal, Dose 1: number analyzed (Participants) | 501 | 503
  Grade 3 Gastrointestinal, Dose 1 | 3 | 2
  Related Gastrointestinal, Dose 1: number analyzed (Participants) | 501 | 503
  Related Gastrointestinal, Dose 1 | 16 | 14
  Any Headache, Dose 1: number analyzed (Participants) | 501 | 503
  Any Headache, Dose 1 | 72 | 42
  Grade 3 Headache, Dose 1: number analyzed (Participants) | 501 | 503
  Grade 3 Headache, Dose 1 | 2 | 4
  Related Headache, Dose 1: number analyzed (Participants) | 501 | 503
  Related Headache, Dose 1 | 58 | 27
  Any Myalgia, Dose 1: number analyzed (Participants) | 501 | 503
  Any Myalgia, Dose 1 | 106 | 27
  Grade 3 Myalgia, Dose 1: number analyzed (Participants) | 501 | 503
  Grade 3 Myalgia, Dose 1 | 6 | 2
  Related Myalgia, Dose 1: number analyzed (Participants) | 501 | 503
  Related Myalgia, Dose 1 | 91 | 16
  Any Shivering, Dose 1: number analyzed (Participants) | 501 | 503
  Any Shivering, Dose 1 | 38 | 17
  Grade 3 Shivering, Dose 1: number analyzed (Participants) | 501 | 503
  Grade 3 Shivering, Dose 1 | 1 | 1
  Related Shivering, Dose 1: number analyzed (Participants) | 501 | 503
  Related Shivering, Dose 1 | 32 | 12
  Any Temperature, Dose 1: number analyzed (Participants) | 501 | 503
  Any Temperature, Dose 1 | 39 | 9
  Grade 3 Temperature, Dose 1: number analyzed (Participants) | 501 | 503
  Grade 3 Temperature, Dose 1 | 0 | 2
  Related Temperature, Dose 1: number analyzed (Participants) | 501 | 503
  Related Temperature, Dose 1 | 31 | 4
  Any Fatigue, Dose 2: number analyzed (Participants) | 492 | 489
  Any Fatigue, Dose 2 | 122 | 39
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 492 | 489
  Grade 3 Fatigue, Dose 2 | 9 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 492 | 489
  Related Fatigue, Dose 2 | 105 | 30
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 492 | 489
  Any Gastrointestinal, Dose 2 | 37 | 19
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 492 | 489
  Grade 3 Gastrointestinal, Dose 2 | 3 | 1
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 492 | 489
  Related Gastrointestinal, Dose 2 | 26 | 13
  Any Headache, Dose 2: number analyzed (Participants) | 492 | 489
  Any Headache, Dose 2 | 76 | 26
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 492 | 489
  Grade 3 Headache, Dose 2 | 4 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 492 | 489
  Related Headache, Dose 2 | 63 | 20
  Any Myalgia, Dose 2: number analyzed (Participants) | 492 | 489
  Any Myalgia, Dose 2 | 113 | 18
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 492 | 489
  Grade 3 Myalgia, Dose 2 | 7 | 0
  Related Myalgia, Dose 2: number analyzed (Participants) | 492 | 489
  Related Myalgia, Dose 2 | 94 | 16
  Any Shivering, Dose 2: number analyzed (Participants) | 492 | 489
  Any Shivering, Dose 2 | 59 | 11
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 492 | 489
  Grade 3 Shivering, Dose 2 | 5 | 1
  Related Shivering, Dose 2: number analyzed (Participants) | 492 | 489
  Related Shivering, Dose 2 | 47 | 9
  Any Temperature, Dose 2: number analyzed (Participants) | 492 | 489
  Any Temperature, Dose 2 | 38 | 6
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 492 | 489
  Grade 3 Temperature, Dose 2 | 0 | 2
  Related Temperature, Dose 2: number analyzed (Participants) | 492 | 489
  Related Temperature, Dose 2 | 35 | 2
  Any Fatigue, Across Doses | 166 | 77
  Grade 3 Fatigue, Across Doses | 16 | 4
  Related Fatigue, Across Doses | 140 | 52
  Any Gastrointestinal, Across Doses | 55 | 40
  Grade 3 Gastrointestinal, Across Doses | 5 | 2
  Related Gastrointestinal, Across Doses | 38 | 21
  Any Headache, Across Doses | 124 | 55
  Grade 3 Headache, Across Doses | 5 | 4
  Related Headache, Across Doses | 104 | 37
  Any Myalgia, Across Doses | 157 | 41
  Grade 3 Myalgia, Across Doses | 12 | 2
  Related Myalgia, Across Doses | 137 | 29
  Any Shivering, Across Doses | 75 | 22
  Grade 3 Shivering, Across Doses | 6 | 2
  Related Shivering, Across Doses | 64 | 16
  Any Temperature, Across Doses | 62 | 13
  Grade 3 Temperature, Across Doses | 0 | 2
  Related Temperature, Across Doses | 54 | 6

14. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Occurrence, intensity and relationship to vaccination of unsolicited AEs during 30 days (Days 0-29) after each vaccination, according to the Medical Dictionary for Regulatory Activities (MedDRA) classification in all subjects. An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within the 30 days (Days 0-29) after each vaccination
Population: This analysis was based on the the total vaccinated cohort, which included all subjects with at least one dose of study vaccine or placebo administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022 GSK1437173A Group | Zoster-022 Placebo Group
Number analyzed (Participants) | 6950 | 6950
Participants
  Any unsolicited AE(s) | 3859 | 2263
  Grade 3 unsolicited AE(s) | 485 | 265
  Related unsolicited AE(s) | 2853 | 529

15. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Month 0 to Month 14
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022 GSK1437173A Group | Zoster-022 Placebo Group
Number analyzed (Participants) | 6950 | 6950
Participants
  Any SAE(s) | 891 | 939
  Related SAE(s) | 12 | 7

16. Secondary Outcome: Number of Subjects With Fatal Serious Adverse Events (SAEs)
Description: as for outcome 15
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022 GSK1437173A Group | Zoster-022 Placebo Group
Number analyzed (Participants) | 6950 | 6950
Participants | 426 | 459

17. Secondary Outcome: Number of Subjects With SAEs Related to Study Participation or Concomitant GSK Medication
Description: The number of subjects with SAEs related to study participation or concomitant GSK medication were tabulated
Time Frame: During the entire study period (3 to 5 year period following day 0)
Population: The analysis was based on the total vaccinated cohort, which included all subjects with at least one dose of study vaccine or placebo administered
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022 GSK1437173A Group | Zoster-022 Placebo Group
Number analyzed (Participants) | 6950 | 6950
Participants | 57 | 84

18. Secondary Outcome: Number of Subjects With Any and Related Potential Immune Mediated Diseases (pIMDs)
Description: Occurrence and relationship to vaccination of any potential immune-mediated diseases (pIMDs) during the entire study period in all subjects
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022 GSK1437173A Group | Zoster-022 Placebo Group
Number analyzed (Participants) | 6950 | 6950
Participants
  Any pIMD | 92 | 97
  Related pIMDs | 8 | 6

19. Secondary Outcome: Number of Subjects With Any and Related Medically Attended Visits
Description: Occurrence and relationship to vaccination of medically attended visits other than routine health care visits, from Month 0 to Month 8 in all subjects. Medically attended visits were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any medically attended visits= Occurrence of any medically attended visits regardless of intensity grade or relation to vaccination.
Time Frame: From Month 0 to Month 8 post-vaccination
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022 GSK1437173A Group | Zoster-022 Placebo Group
Number analyzed (Participants) | 6950 | 6950
Participants
  Any medically attended visits | 2882 | 2911
  Related medically attended visits | 165 | 66

20. Secondary Outcome: Outcome Measure for the Pooled Analysis of Combined Data From Studies Zoster-006 (NCT01165177) and Zoster-022 (NCT01165229): Overall Number of Subjects With PHN in Subjects ≥ 50 YOA
Description: Incidence of PHN calculated using the mTVc during the entire study period in subjects ≥ 50 YOA.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Zoster-022/006 Pooled GSK1437173A 50-59 YOA Group: Subjects between 50 and 59 years of age (YOA), receiving herpes zoster subunit vaccine (gE/AS01B vaccine) according to a 0, 2-month schedule.
- Zoster-022/006 Pooled GSK1437173A 60-69 YOA Group: Subjects between 60 and 69 years of age (YOA), receiving herpes zoster subunit vaccine (gE/AS01B vaccine) according to a 0, 2-month schedule.
- Zoster-022/006 Pooled GSK1437173A 70-79 YOA Group: Subjects between 70 and 79 years of age (YOA), receiving herpes zoster subunit vaccine (gE/AS01B vaccine) according to a 0, 2-month schedule.
- Zoster-022/006 Pooled GSK1437173A >=80 YOA Group: Subjects above 80 years of age (YOA), receiving herpes zoster subunit vaccine (gE/AS01B vaccine) according to a 0, 2-month schedule.
- Zoster-022/006 Pooled GSK1437173A >=50 YOA Group: Subjects above 50 years of age (YOA), receiving herpes zoster subunit vaccine (gE/AS01B vaccine) according to a 0, 2-month schedule.
- Zoster-022/006 Pooled Placebo 50-59 YOA Group: Subjects between 50 and 59 years of age (YOA), receiving saline solution (NaCl solution) as control according to a 0, 2-month schedule.
- Zoster-022/006 Pooled Placebo 60-69 YOA Group: Subjects between 60 and 69 years of age (YOA), receiving saline solution (NaCl solution) as control according to a 0, 2-month schedule.
- Zoster-022/006 Pooled Placebo 70-79 YOA Group: Subjects between 70 and 79 years of age (YOA), receiving saline solution (NaCl solution) as control according to a 0, 2-month schedule.
- Zoster-022/006 Pooled Placebo >=80 YOA Group: Subjects above 80 years of age (YOA), receiving saline solution (NaCl solution) as control according to a 0, 2-month schedule.
- Zoster-022/006 Pooled Placebo >=50 YOA Group: Subjects above 50 years of age (YOA), receiving saline solution (NaCl solution) as control according to a 0, 2-month schedule.
Arm/Group | Zoster-022/006 Pooled GSK1437173A 50-59 YOA Group | Zoster-022/006 Pooled GSK1437173A 60-69 YOA Group | Zoster-022/006 Pooled GSK1437173A 70-79 YOA Group | Zoster-022/006 Pooled GSK1437173A >=80 YOA Group | Zoster-022/006 Pooled GSK1437173A >=50 YOA Group | Zoster-022/006 Pooled Placebo 50-59 YOA Group | Zoster-022/006 Pooled Placebo 60-69 YOA Group | Zoster-022/006 Pooled Placebo 70-79 YOA Group | Zoster-022/006 Pooled Placebo >=80 YOA Group | Zoster-022/006 Pooled Placebo >=50 YOA Group
Number analyzed (Participants) | 3491 | 2140 | 6468 | 1782 | 13881 | 3523 | 2166 | 6554 | 1792 | 14035
Participants | 0 | 0 | 2 | 2 | 4 | 8 | 2 | 29 | 7 | 46
Statistical Analysis 1: Comparison: Zoster-022/006 Pooled GSK1437173A 50-59 YOA Group vs Zoster-022/006 Pooled Placebo 50-59 YOA Group; Comparison of vaccine efficacy in prevention of PHN between Zoster-022/006 Pooled GSK1437173A 50-59YOA Group and Zoster-022/006 Pooled Placebo 50-59YOA Group.Comparison of vaccine efficacy for groups 70-79 and above 80 YOA are presented in outcome measure 2; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0081, Poisson exact test; Vaccine efficacy = 100.00, 95% CI 2-sided [40.88 to 100.00]
Statistical Analysis 2: Comparison: Zoster-022/006 Pooled GSK1437173A 60-69 YOA Group vs Zoster-022/006 Pooled Placebo 60-69 YOA Group; Comparison of vaccine efficacy in prevention of PHN between Zoster-022/006 Pooled GSK1437173A 60-69YOA Group and Zoster-022/006 Pooled Placebo 60-69YOA Group; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.5097, Poisson exact test; Vaccine efficacy = 100.00, 95% CI 2-sided [-442.83 to 100.00]

21. Secondary Outcome: Outcome Measure for the Pooled Analysis of Combined Data From Studies Zoster-006 (NCT01165177) and Zoster-022 (NCT01165229): Number of Subjects With a Reduction of PHN Incidence in Subjects ≥ 50 YOA With Confirmed HZ
Description: Occurrence of PHN during the entire study period in all subjects with confirmed HZ.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022/006 Pooled GSK1437173A 50-59 YOA Group | Zoster-022/006 Pooled GSK1437173A 60-69 YOA Group | Zoster-022/006 Pooled GSK1437173A 70-79 YOA Group | Zoster-022/006 Pooled GSK1437173A >=80 YOA Group | Zoster-022/006 Pooled GSK1437173A >=50 YOA Group | Zoster-022/006 Pooled Placebo 50-59 YOA Group | Zoster-022/006 Pooled Placebo 60-69 YOA Group | Zoster-022/006 Pooled Placebo 70-79 YOA Group | Zoster-022/006 Pooled Placebo >=80 YOA Group | Zoster-022/006 Pooled Placebo >=50 YOA Group
Number analyzed (Participants) | 4 | 3 | 19 | 6 | 32 | 103 | 90 | 216 | 68 | 477
Participants | 0 | 0 | 2 | 2 | 4 | 8 | 2 | 29 | 7 | 46
Statistical Analysis 1: Comparison: Zoster-022/006 Pooled GSK1437173A 50-59 YOA Group vs Zoster-022/006 Pooled Placebo 50-59 YOA Group; Comparison of Vaccine efficacy in reduction of PHN incidence in subjects with confirmed HZ episode in Zoster-022/006 Pooled GSK1437173A 50-59 YOA Group versus Zoster-022/006 Pooled Placebo 50-59 YOA Group; Test type: Other — The efficacy of HZ/su vaccine in reduction of PHN in subjects with confirmed HZ episodes was demonstrated if the LL of the two-sided 95% CI of VE was above 0%; p = 1.0000, Poisson exact test; Vaccine efficacy = 100.00, 95% CI 2-sided [-649.86 to 100.00]
Statistical Analysis 2: Comparison: Zoster-022/006 Pooled GSK1437173A 60-69 YOA Group vs Zoster-022/006 Pooled Placebo 60-69 YOA Group; Comparison of Vaccine efficacy in reduction of PHN incidence in subjects with confirmed HZ episode in Zoster-022/006 Pooled GSK1437173A 60-69 YOA Group versus Zoster-022/006 Pooled Placebo 60-69 YOA Group; Test type: Other — [test comment as in outcome 21, analysis 1]; p = 1.0000, Poisson exact test; Vaccine efficacy = 100.00, 95% CI 2-sided [-3938.70 to 100.00]
Statistical Analysis 3: Comparison: Zoster-022/006 Pooled GSK1437173A 70-79 YOA Group vs Zoster-022/006 Pooled Placebo 70-79 YOA Group; Comparison of Vaccine efficacy in reduction of PHN incidence in subjects with confirmed HZ episode in Zoster-022/006 Pooled GSK1437173A 70-79 YOA Group versus Zoster-022/006 Pooled Placebo 70-79 YOA Group; Test type: Other — [test comment as in outcome 21, analysis 1]; p = 1.0000, Poisson exact test; Vaccine efficacy = 21.60, 95% CI 2-sided [-149.41 to 78.91]
Statistical Analysis 4: Comparison: Zoster-022/006 Pooled GSK1437173A >=80 YOA Group vs Zoster-022/006 Pooled Placebo >=80 YOA Group; Comparison of Vaccine efficacy in reduction of PHN incidence in subjects with confirmed HZ episode in Zoster-022/006 Pooled GSK1437173A >=80 YOA Group versus Zoster-022/006 Pooled Placebo>=80 YOA Group; Test type: Other — [test comment as in outcome 21, analysis 1]; p = 0.1528, Poisson exact test; Vaccine efficacy = -223.81, 95% CI 2-sided [-883.05 to 18.84]
Statistical Analysis 5: Comparison: Zoster-022/006 Pooled GSK1437173A >=50 YOA Group vs Zoster-022/006 Pooled Placebo >=50 YOA Group; Comparison of Vaccine efficacy in reduction of PHN incidence in subjects with confirmed HZ episode in Zoster-022/006 Pooled GSK1437173A >=50 YOA Group versus Zoster-022/006 Pooled Placebo >=50 YOA Group; Test type: Other — [test comment as in outcome 21, analysis 1]; p = 0.5417, Poisson exact test; Vaccine efficacy = 0.29, 95% CI 2-sided [-161.53 to 65.57]

22. Secondary Outcome: Outcome Measure for the Pooled Analysis of Combined Data From Studies Zoster-006 (NCT01165177) and Zoster-022 (NCT01165229): Number of Subjects With at Least One Day of Severe 'Worst' HZ-associated Pain in Subjects ≥ 70 YOA With Confirmed HZ.
Description: The duration of severe 'worst' HZ-associated pain following the onset of a confirmed HZ rash over the entire pain reporting period was measured by the ZBPI in subjects ≥ 70 YOA with confirmed HZ .
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Zoster-022/006 Pooled GSK1437173A >=70 YOA Group: Subjects above 70 years of age (YOA), receiving herpes zoster subunit vaccine (gE/AS01B vaccine) according to a 0, 2-month schedule.
- Zoster-022/006 Pooled Placebo >=70 YOA Group: Subjects above 70 years of age (YOA), receiving saline solution (NaCl solution) as control according to a 0, 2-month schedule.
Arm/Group | Zoster-022/006 Pooled GSK1437173A 70-79 YOA Group | Zoster-022/006 Pooled GSK1437173A >=80 YOA Group | Zoster-022/006 Pooled GSK1437173A >=70 YOA Group | Zoster-022/006 Pooled Placebo 70-79 YOA Group | Zoster-022/006 Pooled Placebo >=80 YOA Group | Zoster-022/006 Pooled Placebo >=70 YOA Group
Number analyzed (Participants) | 19 | 6 | 25 | 216 | 68 | 284
Participants | 17 | 3 | 20 | 193 | 61 | 254
Statistical Analysis 1: Comparison: Zoster-022/006 Pooled GSK1437173A 70-79 YOA Group vs Zoster-022/006 Pooled Placebo 70-79 YOA Group; Comparison of VE in reduction of duration of severe worst HZ associated pain between Zoster-022/006 pooled GSK1437173A 70-79YOA Group and Zoster-022/006 pooled Placebo 70-79YOA Group; Test type: Other — The VE of HZ/su against duration of severe worst pain in subjects with confirmed HZ was demonstrated if the LL of the two-sided 95% CI of VE derived from the Hazard ratio was above 0%; p = 0.2885, Poisson exact test; Vaccine efficacy = 23.75, 95% CI 2-sided [-25.80 to 53.78]
Statistical Analysis 2: Comparison: Zoster-022/006 Pooled GSK1437173A >=80 YOA Group vs Zoster-022/006 Pooled Placebo >=80 YOA Group; Comparison of VE in reduction of duration of severe worst HZ associated pain between Zoster-022/006 pooled GSK1437173A >=80 YOA Group and Zoster-022/006 pooled Placebo >=80 YOA Group; Test type: Other — [test comment as in outcome 22, analysis 1]; p = 0.1940, Poisson exact test; Vaccine efficacy = 54.93, 95% CI 2-sided [-50.03 to 86.46]
Statistical Analysis 3: Comparison: Zoster-022/006 Pooled GSK1437173A >=70 YOA Group vs Zoster-022/006 Pooled Placebo >=70 YOA Group; Comparison of VE in reduction of duration of severe worst HZ associated pain between Zoster-022/006 pooled GSK1437173A >=70 YOA Group and Zoster-022/006 pooled Placebo>=70 YOA Group; Test type: Other — [test comment as in outcome 22, analysis 1]; p = 0.1243, Poisson exact test; Vaccine efficacy = 30.48, 95% CI 2-sided [-10.52 to 56.27]

23. Secondary Outcome: Outcome Measure for the Pooled Analysis of Combined Data From Studies Zoster-006 (NCT01165177) and Zoster-022 (NCT01165229): Duration of Severe 'Worst' HZ-associated Pain in Subjects ≥ 70 YOA With Confirmed HZ.
Description: Duration of severe 'worst' HZ-associated pain following the onset of a confirmed HZ rash over the entire pain reporting period was measured by the ZBPI in subjects ≥ 70 YOA with confirmed HZ.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Zoster-022/006 Pooled GSK1437173A 70-79 YOA Group | Zoster-022/006 Pooled GSK1437173A >=80 YOA Group | Zoster-022/006 Pooled GSK1437173A >=70 YOA Group | Zoster-022/006 Pooled Placebo 70-79 YOA Group | Zoster-022/006 Pooled Placebo >=80 YOA Group | Zoster-022/006 Pooled Placebo >=70 YOA Group
Number analyzed (Participants) | 17 | 3 | 20 | 193 | 61 | 254
Days | 20.3 (29.71) | 98.7 (57.73) | 32.1 (43.80) | 48.3 (96.34) | 45.2 (95.58) | 47.5 (95.98)

24. Secondary Outcome: Outcome Measure for the Pooled Analysis of Combined Data From Studies Zoster-006 (NCT01165177) and Zoster-022 (NCT01165229): Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Occurrence, intensity of each solicited local symptom within 7 days (Days 0-6) after each vaccination, in subjects ≥ 70 YOA. Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: Within the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Groups:
- Zoster-022/006 Pooled GSK1437173A Group: Subjects receiving herpes zoster subunit vaccine (gE/AS01B vaccine) according to a 0, 2-month schedule.
- Zoster-022/006 Pooled Placebo Group: Subjects receiving saline solution (NaCl solution) as control according to a 0, 2-month schedule.
Arm/Group | Zoster-022/006 Pooled GSK1437173A Group | Zoster-022/006 Pooled Placebo Group
Number analyzed (Participants) | 2258 | 2263
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 2246 | 2255
  Any Pain, Dose 1 | 1336 | 128
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 2246 | 2255
  Grade 3 Pain, Dose 1 | 42 | 1
  Any Redness, Dose 1: number analyzed (Participants) | 2246 | 2255
  Any Redness, Dose 1 | 606 | 17
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 2246 | 2255
  Grade 3 Redness, Dose 1 | 43 | 0
  Any Swelling, Dose 1: number analyzed (Participants) | 2246 | 2255
  Any Swelling, Dose 1 | 355 | 17
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 2246 | 2255
  Grade 3 Swelling, Dose 1 | 17 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 2160 | 2169
  Any Pain, Dose 2 | 1241 | 107
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 2160 | 2169
  Grade 3 Pain, Dose 2 | 60 | 3
  Any Redness, Dose 2: number analyzed (Participants) | 2160 | 2169
  Any Redness, Dose 2 | 582 | 14
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 2160 | 2169
  Grade 3 Redness, Dose 2 | 39 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 2160 | 2169
  Any Swelling, Dose 2 | 344 | 10
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 2160 | 2169
  Grade 3 Swelling, Dose 2 | 15 | 0
  Any Pain, Across Doses | 1562 | 199
  Grade 3 Pain, Across Doses | 90 | 4
  Any Redness, Across Doses | 851 | 27
  Grade 3 Redness, Across Doses | 70 | 0
  Any Swelling, Across Doses | 519 | 25
  Grade 3 Swelling, Across Doses | 30 | 0

25. Secondary Outcome: Outcome Measure for the Pooled Analysis of Combined Data From Studies Zoster-006 (NCT01165177) and Zoster-022 (NCT01165229): Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache, myalgia, shivering and fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = Temperature> 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022/006 Pooled GSK1437173A Group | Zoster-022/006 Pooled Placebo Group
Number analyzed (Participants) | 2252 | 2264
Participants
  Any Fatigue, Dose 1: number analyzed (Participants) | 2237 | 2256
  Any Fatigue, Dose 1 | 545 | 231
  Grade 3 Fatigue, Dose 1: number analyzed (Participants) | 2237 | 2256
  Grade 3 Fatigue, Dose 1 | 31 | 13
  Related Fatigue, Dose 1: number analyzed (Participants) | 2237 | 2256
  Related Fatigue, Dose 1 | 441 | 147
  Any Gastrointestinal, Dose 1: number analyzed (Participants) | 2237 | 2256
  Any Gastrointestinal, Dose 1 | 170 | 123
  Grade 3 Gastrointestinal, Dose 1: number analyzed (Participants) | 2237 | 2256
  Grade 3 Gastrointestinal, Dose 1 | 15 | 6
  Related Gastrointestinal, Dose 1: number analyzed (Participants) | 2237 | 2256
  Related Gastrointestinal, Dose 1 | 101 | 67
  Any Headache, Dose 1: number analyzed (Participants) | 2237 | 2256
  Any Headache, Dose 1 | 380 | 189
  Grade 3 Headache, Dose 1: number analyzed (Participants) | 2237 | 2256
  Grade 3 Headache, Dose 1 | 7 | 8
  Related Headache, Dose 1: number analyzed (Participants) | 2237 | 2256
  Related Headache, Dose 1 | 293 | 132
  Any Myalgia, Dose 1: number analyzed (Participants) | 2237 | 2256
  Any Myalgia, Dose 1 | 530 | 159
  Grade 3 Myalgia, Dose 1: number analyzed (Participants) | 2237 | 2256
  Grade 3 Myalgia, Dose 1 | 26 | 7
  Related Myalgia, Dose 1: number analyzed (Participants) | 2237 | 2256
  Related Myalgia, Dose 1 | 445 | 101
  Any Shivering, Dose 1: number analyzed (Participants) | 2237 | 2256
  Any Shivering, Dose 1 | 206 | 73
  Grade 3 Shivering, Dose 1: number analyzed (Participants) | 2237 | 2256
  Grade 3 Shivering, Dose 1 | 15 | 3
  Related Shivering, Dose 1: number analyzed (Participants) | 2237 | 2256
  Related Shivering, Dose 1 | 173 | 50
  Any Temperature, Dose 1: number analyzed (Participants) | 2237 | 2256
  Any Temperature, Dose 1 | 142 | 34
  Grade 3 Temperature, Dose 1: number analyzed (Participants) | 2237 | 2256
  Grade 3 Temperature, Dose 1 | 1 | 2
  Related Temperature, Dose 1: number analyzed (Participants) | 2237 | 2256
  Related Temperature, Dose 1 | 111 | 16
  Any Fatigue, Dose 2: number analyzed (Participants) | 2159 | 2166
  Any Fatigue, Dose 2 | 579 | 169
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 2159 | 2166
  Grade 3 Fatigue, Dose 2 | 53 | 4
  Related Fatigue, Dose 2: number analyzed (Participants) | 2159 | 2166
  Related Fatigue, Dose 2 | 495 | 116
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 2159 | 2166
  Any Gastrointestinal, Dose 2 | 188 | 75
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 2159 | 2166
  Grade 3 Gastrointestinal, Dose 2 | 14 | 5
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 2159 | 2166
  Related Gastrointestinal, Dose 2 | 142 | 35
  Any Headache, Dose 2: number analyzed (Participants) | 2159 | 2166
  Any Headache, Dose 2 | 455 | 133
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 2159 | 2166
  Grade 3 Headache, Dose 2 | 30 | 2
  Related Headache, Dose 2: number analyzed (Participants) | 2159 | 2166
  Related Headache, Dose 2 | 386 | 86
  Any Myalgia, Dose 2: number analyzed (Participants) | 2159 | 2166
  Any Myalgia, Dose 2 | 560 | 112
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 2159 | 2166
  Grade 3 Myalgia, Dose 2 | 42 | 4
  Related Myalgia, Dose 2: number analyzed (Participants) | 2159 | 2166
  Related Myalgia, Dose 2 | 484 | 75
  Any Shivering, Dose 2: number analyzed (Participants) | 2159 | 2166
  Any Shivering, Dose 2 | 334 | 55
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 2159 | 2166
  Grade 3 Shivering, Dose 2 | 36 | 4
  Related Shivering, Dose 2: number analyzed (Participants) | 2159 | 2166
  Related Shivering, Dose 2 | 292 | 34
  Any Temperature, Dose 2: number analyzed (Participants) | 2159 | 2166
  Any Temperature, Dose 2 | 224 | 30
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 2159 | 2166
  Grade 3 Temperature, Dose 2 | 2 | 3
  Related Temperature, Dose 2: number analyzed (Participants) | 2159 | 2166
  Related Temperature, Dose 2 | 189 | 14
  Any Fatigue, Across Doses | 825 | 326
  Grade 3 Fatigue, Across Doses | 79 | 17
  Related Fatigue, Across Doses | 699 | 220
  Any Gastrointestinal, Across Doses | 304 | 172
  Grade 3 Gastrointestinal,Across Doses | 26 | 10
  Related Gastrointestinal,Across Doses | 210 | 91
  Any Headache, Across Doses | 653 | 268
  Grade 3 Headache, Across Doses | 34 | 10
  Related Headache, Across Doses | 547 | 185
  Any Myalgia, Across Doses | 790 | 225
  Grade 3 Myalgia, Across Doses | 62 | 10
  Related Myalgia, Across Doses | 689 | 157
  Any Shivering, Across Doses | 439 | 110
  Grade 3 Shivering, Across Doses | 49 | 6
  Related Shivering, Across Doses | 380 | 75
  Any Temperature, Across Doses | 323 | 61
  Grade 3 Temperature, Across Doses | 3 | 3
  Related Temperature, Across Doses | 265 | 30

26. Secondary Outcome: Outcome Measure for the Pooled Analysis of Combined Data From Studies Zoster-006 (NCT01165177) and Zoster-022 (NCT01165229): Number of Subjects With Any,Grade 3 and Related Unsolicited AEs in Subjects ≥ 70 YOA
Description: Occurrence, intensity and relationship to vaccination of unsolicited AEs during 30 days (Days 0-29) after each vaccination, according to the MedDRA classification, in subjects ≥ 70 YOA.An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within 30 days (Days 0 - 29) after each vaccination
Population: The analysis was based on the total vaccinated cohort, which included all vaccinated subjects with study vaccine or placebo administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022/006 Pooled GSK1437173A Group | Zoster-022/006 Pooled Placebo Group
Number analyzed (Participants) | 8758 | 8773
Participants
  Any unsolicited AE(s) | 4366 | 2732
  Grade 3 unsolicited AE(s) | 553 | 335
  Related unsolicited AE(s) | 2961 | 578

27. Secondary Outcome: Outcome Measure for the Pooled Analysis of Combined Data From Studies Zoster-006 (NCT01165177) and Zoster-022 (NCT01165229): Number of Subjects With Any and Related SAEs
Description: Occurrence and relationship to vaccination of all SAEs from Month 0 to Month 14 in subjects ≥ 70 YOA. Related SAEs also included any SAEs related to study participation or concurrent GSK medication/vaccine.
Time Frame: From Month 0 to Month 14
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022/006 Pooled GSK1437173A Group | Zoster-022/006 Pooled Placebo Group
Number analyzed (Participants) | 8758 | 8773
Participants
  Any SAE(s) | 1117 | 1171
  Related SAE(s) | 12 | 7

28. Secondary Outcome: Outcome Measure for the Pooled Analysis of Combined Data From Studies Zoster-006 (NCT01165177) and Zoster-022 (NCT01165229): Number of Subjects With Fatal SAEs
Description: Fatal SAEs during the entire study period in subjects ≥ 70 YOA.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022/006 Pooled GSK1437173A Group | Zoster-022/006 Pooled Placebo Group
Number analyzed (Participants) | 8758 | 8773
Participants | 128 | 144

29. Secondary Outcome: Outcome Measure for the Pooled Analysis of Combined Data From Studies Zoster-006 (NCT01165177) and Zoster-022 (NCT01165229): Number of Subjects With Any and Related pIMDs
Description: Occurrence and relationship to vaccination of any pIMDs during the entire study period in subjects ≥ 70 YOA.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022/006 Pooled GSK1437173A Group | Zoster-022/006 Pooled Placebo Group
Number analyzed (Participants) | 8758 | 8773
Participants
  Any pIMD(s) | 110 | 118
  Related pIMD(s) | 8 | 8

30. Secondary Outcome: Outcome Measure for the Pooled Analysis of Combined Data From Studies Zoster-006 (NCT01165177) and Zoster-022 (NCT01165229): Number of Subjects With Any and Related Medically Attended Visits
Description: Occurrence and relationship to vaccination of medically attended visits (defined as hospitalizations, emergency room visits or visits to or from medical personnel), other than routine health care visits, from Month 0 to Month 8 in subjects ≥ 70 YOA.
Time Frame: From Month 0 to Month 8 post-vaccination
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster-022/006 Pooled GSK1437173A Group | Zoster-022/006 Pooled Placebo Group
Number analyzed (Participants) | 8758 | 8773
Participants
  Any medically attended visits | 3593 | 3648
  Related medically attended visits | 180 | 80

ADVERSE EVENTS:
Time Frame: Solicited symptoms: within 7 days (Days 0-6) after vaccination; Unsolicited adverse events: within 30 days (Days 0-29) after vaccination; Serious Adverse Events (SAEs): during the entire study period (3 to 5 year period following Day 0).
Arm/Group | Zoster-022 GSK1437173A Group | Zoster-022 Placebo Group
All-Cause Mortality (participants affected / at risk) | 426/6950 | 459/6950
Serious Adverse Events (participants affected / at risk) | 1153/6950 | 1214/6950
Other Adverse Events (participants affected / at risk) | 3067/6950 | 610/6950
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoster-022 GSK1437173A Group (N=6950) | Zoster-022 Placebo Group (N=6950)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 13 (15)
Anaemia vitamin b12 deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hypersplenism (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pernicious anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Acute coronary syndrome (Cardiac disorders) | 3 (3) | 4 (6)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 21 (22) | 28 (29)
Angina pectoris (Cardiac disorders) | 13 (13) | 6 (6)
Angina unstable (Cardiac disorders) | 7 (7) | 7 (7)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 3 (3)
Arrhythmia (Cardiac disorders) | 5 (5) | 9 (9)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 40 (45) | 54 (56)
Atrial flutter (Cardiac disorders) | 6 (6) | 5 (5)
Atrioventricular block (Cardiac disorders) | 0 (0) | 4 (4)
Atrioventricular block complete (Cardiac disorders) | 4 (4) | 2 (2)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 3 (3)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 4 (4) | 8 (8)
Cardiac arrest (Cardiac disorders) | 23 (23) | 17 (17)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 51 (52) | 57 (62)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 3 (3) | 6 (6)
Cardiac failure congestive (Cardiac disorders) | 23 (23) | 33 (37)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 2 (2) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 5 (5)
Cardiogenic shock (Cardiac disorders) | 6 (6) | 2 (2)
Cardiomegaly (Cardiac disorders) | 0 (0) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 2 (2)
Chronotropic incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 2 (2) | 1 (1)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 28 (29) | 25 (25)
Coronary artery insufficiency (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 3 (3) | 6 (6)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Heart valve incompetence (Cardiac disorders) | 0 (0) | 2 (2)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 4 (4)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 3 (3)
Myocardial infarction (Cardiac disorders) | 41 (43) | 45 (45)
Myocardial ischaemia (Cardiac disorders) | 5 (6) | 16 (16)
Palpitations (Cardiac disorders) | 1 (1) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 2 (2) | 1 (1)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 5 (5) | 6 (6)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3) | 2 (2)
Tricuspid valve incompetence (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 6 (8)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Renal dysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 4 (4)
Vertigo positional (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 3 (3)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 1 (1)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 3 (3)
Age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 7 (7) | 7 (7)
Choroidal effusion (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Iridocele (Eye disorders) | 1 (1) | 0 (0)
Iritis (Eye disorders) | 0 (0) | 1 (1)
Ocular hypertension (Eye disorders) | 0 (0) | 1 (1)
Ocular vascular disorder (Eye disorders) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 2 (2) | 0 (0)
Retinal degeneration (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 4 (4)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 3 (3) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diaphragmatic hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Diverticulum (Gastrointestinal disorders) | 3 (3) | 3 (3)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 4 (4) | 6 (6)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 4 (4)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 6 (6)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 4 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 6 (6) | 7 (7)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 5 (5) | 10 (10)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 6 (6) | 6 (6)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Large intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 3 (3) | 4 (4)
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 (1) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric artery embolism (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 8 (8)
Pancreatitis acute (Gastrointestinal disorders) | 5 (5) | 4 (5)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 4 (4)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Accidental death (General disorders) | 1 (1) | 0 (0)
Administration site erythema (General disorders) | 1 (1) | 0 (0)
Administration site pain (General disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Cardiac death (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 3 (4)
Chest pain (General disorders) | 20 (20) | 19 (20)
Chills (General disorders) | 1 (1) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 17 (17) | 29 (29)
Device battery issue (General disorders) | 0 (0) | 1 (1)
Device deposit issue (General disorders) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 1 (1) | 2 (2)
Device leakage (General disorders) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 1 (1)
Drowning (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 2 (2)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Ill-defined disorder (General disorders) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 1 (1) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 9 (9) | 12 (12)
Non-cardiac chest pain (General disorders) | 0 (0) | 4 (4)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Organ failure (General disorders) | 2 (2) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Sudden cardiac death (General disorders) | 2 (2) | 3 (3)
Sudden death (General disorders) | 13 (13) | 4 (4)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 1 (1)
Thrombosis in device (General disorders) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 3 (3) | 3 (3)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 5 (5) | 5 (5)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 7 (8) | 15 (17)
Cholecystitis acute (Hepatobiliary disorders) | 7 (7) | 4 (4)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 14 (14) | 14 (14)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chronic hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder perforation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Allergic granulomatous angiitis (Immune system disorders) | 1 (1) | 0 (0)
Amyloidosis (Immune system disorders) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Abdominal abscess (Infections and infestations) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Alcaligenes infection (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Anal fistula infection (Infections and infestations) | 0 (0) | 1 (1)
Anorectal cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 5 (5) | 5 (5)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Arteriosclerotic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 2 (2)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 2 (2) | 2 (2)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 8 (8) | 7 (8)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 4 (4)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Candida sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cavernous sinus thrombosis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 8 (8) | 14 (14)
Cholecystitis infective (Infections and infestations) | 1 (1) | 1 (1)
Clostridium bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 5 (5)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1)
Colonic abscess (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 4 (4) | 0 (0)
Cystitis klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (1)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 5 (5) | 11 (11)
Empyema (Infections and infestations) | 1 (1) | 2 (2)
Encephalitis (Infections and infestations) | 1 (1) | 1 (1)
Encephalitis viral (Infections and infestations) | 1 (1) | 1 (1)
Endocarditis (Infections and infestations) | 3 (3) | 0 (0)
Enterocolitis viral (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 3 (4) | 7 (7)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 8 (8) | 8 (8)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 2 (2)
Graft infection (Infections and infestations) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 3 (3)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster meningitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster oticus (Infections and infestations) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Infectious colitis (Infections and infestations) | 1 (1) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Intestinal gangrene (Infections and infestations) | 2 (2) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1) | 1 (1)
Liver abscess (Infections and infestations) | 2 (2) | 1 (1)
Lobar pneumonia (Infections and infestations) | 4 (4) | 8 (8)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 2 (2)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 1 (1)
Necrotising fasciitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Neuroborreliosis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 2 (2)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 3 (3)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Ovarian abscess (Infections and infestations) | 0 (0) | 1 (1)
Pancreatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 4 (4) | 4 (4)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 70 (73) | 81 (86)
Pneumonia bacterial (Infections and infestations) | 3 (4) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 3 (3)
Postoperative abscess (Infections and infestations) | 3 (3) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 2 (2)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Psittacosis (Infections and infestations) | 1 (1) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Purulence (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 3 (3) | 4 (4)
Pyelonephritis acute (Infections and infestations) | 4 (4) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory moniliasis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 26 (27) | 17 (17)
Septic shock (Infections and infestations) | 11 (11) | 14 (14)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 4 (4) | 1 (1)
Staphylococcal osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 2 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 28 (32) | 24 (27)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 7 (8) | 9 (9)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 3 (3)
Viral infection (Infections and infestations) | 2 (2) | 2 (2)
Vulvitis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 3 (3) | 2 (2)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Back injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Bone fissure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye penetration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 8 (8) | 5 (5)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Femur fracture (Injury, poisoning and procedural complications) | 10 (10) | 15 (15)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Hip fracture (Injury, poisoning and procedural complications) | 7 (7) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Kidney contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Radius fracture (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 6 (6) | 7 (7)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 6 (6) | 1 (1)
Spinal cord injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 9 (10) | 6 (6)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Toxicity to various agents (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood glucose fluctuation (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 8 (8) | 8 (8)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (6) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Marasmus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 5 (5) | 6 (6)
Uraemic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 26 (26) | 17 (17)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Still's disease adult onset (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Acral lentiginous melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute monocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenal gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anaplastic thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 13 (13)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Central nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 6 (6)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large b-cell lymphoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 6 (6)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 1 (1)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Large cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 6 (6)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung adenocarcinoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 4 (4)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 (23) | 13 (13)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 3 (3)
Malignant fibrous histiocytoma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant lymphoma unclassifiable high grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant mast cell neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant neoplasm of ampulla of vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Metastases to gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 5 (5)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Metastases to stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Non-small cell lung cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 10 (10)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Paraganglion neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (19) | 18 (18)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Prostate cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urethral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 2 (2) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 2 (2)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Basilar artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Carotid sinus syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Cerebellar ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral artery thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 6 (6) | 7 (7)
Cerebral infarction (Nervous system disorders) | 16 (16) | 17 (17)
Cerebral ischaemia (Nervous system disorders) | 2 (2) | 3 (3)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 34 (34) | 31 (33)
Cerebrovascular disorder (Nervous system disorders) | 3 (3) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 4 (4) | 2 (2)
Dementia alzheimer's type (Nervous system disorders) | 2 (2) | 0 (0)
Dementia with lewy bodies (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic coma (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 5 (5)
Drop attacks (Nervous system disorders) | 0 (0) | 1 (1)
Dural arteriovenous fistula (Nervous system disorders) | 0 (0) | 1 (1)
Dyspraxia (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 4 (4)
Generalised tonic-clonic seizure (Nervous system disorders) | 2 (2) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 1 (1) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 1 (1)
Hypertonia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 7 (7) | 6 (6)
Lacunar infarction (Nervous system disorders) | 2 (2) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Miller fisher syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Mixed dementia (Nervous system disorders) | 1 (1) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 2 (2)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 2 (2)
Progressive supranuclear palsy (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 4 (4) | 4 (4)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Senile dementia (Nervous system disorders) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 5 (5) | 7 (7)
Syncope (Nervous system disorders) | 11 (11) | 20 (22)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Thrombotic cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Transient global amnesia (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 20 (22) | 14 (15)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Viiith nerve lesion (Nervous system disorders) | 1 (1) | 0 (0)
Viith nerve paralysis (Nervous system disorders) | 2 (2) | 2 (2)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Breathing-related sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 3 (3)
Depressed mood (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 3 (3)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 2 (2)
Major depression (Psychiatric disorders) | 0 (0) | 2 (2)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 2 (2)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizoaffective disorder bipolar type (Psychiatric disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1)
Somatoform disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 18 (19) | 19 (20)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 2 (2)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 4 (4) | 11 (12)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis interstitial (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephroangiosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 6 (6) | 2 (2)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal cyst (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 11 (11) | 11 (12)
Renal hypertension (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 4 (4)
Urethral haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral meatus stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 2 (2) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (3) | 3 (3)
Urinary tract disorder (Renal and urinary disorders) | 1 (1) | 1 (1)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 9 (9) | 7 (7)
Breast dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 4 (4)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal ulceration (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 21 (26) | 18 (18)
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 8 (8)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 21 (21)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 15 (15)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Rectal polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aneurysm ruptured (Vascular disorders) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 6 (6) | 2 (2)
Aortic aneurysm rupture (Vascular disorders) | 4 (4) | 4 (4)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 2 (2)
Aortic occlusion (Vascular disorders) | 1 (1) | 0 (0)
Aortic rupture (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 8 (8)
Arteriosclerosis (Vascular disorders) | 1 (1) | 5 (7)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 5 (5) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 6 (6) | 9 (10)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
Femoral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 6 (6)
Haemorrhage (Vascular disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 22 (22) | 25 (27)
Hypertensive crisis (Vascular disorders) | 7 (8) | 6 (6)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 6 (6) | 5 (5)
Inferior vena caval occlusion (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 0 (0) | 2 (2)
Internal haemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Labile hypertension (Vascular disorders) | 1 (1) | 0 (0)
Microscopic polyangiitis (Vascular disorders) | 0 (0) | 1 (1)
Necrosis ischaemic (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 4 (4)
Peripheral arterial occlusive disease (Vascular disorders) | 6 (6) | 6 (6)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Temporal arteritis (Vascular disorders) | 1 (1) | 1 (1)
Thromboangiitis obliterans (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoster-022 GSK1437173A Group (N=6950) | Zoster-022 Placebo Group (N=6950)
Chills (General disorders) | 353 (415) | 39 (46)
Fatigue (General disorders) | 474 (592) | 169 (192)
Headache (Nervous system disorders) | 586 (717) | 243 (307)
Injection site erythema (General disorders) | 864 (1150) | 27 (29)
Injection site pain (General disorders) | 1975 (2762) | 148 (165)
Injection site swelling (General disorders) | 613 (773) | 16 (18)
Myalgia (Musculoskeletal and connective tissue disorders) | 378 (472) | 99 (113)
Pain (General disorders) | 428 (669) | 60 (67)
Pyrexia (General disorders) | 535 (633) | 52 (56)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.